CLINICAL TRIAL: NCT02227680
Title: Massage Therapy vs. Music Therapy vs. Usual Care in an Inpatient Setting: A Pilot Study
Brief Title: Massage Therapy Versus Music Therapy Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Muscular Therapy Institute Foundation, Inc. (Other); Berklee College of Music (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-32796
Record Dates: First submitted 2014-08-21; First posted 2014-08-28 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: ALL
Keywords: music therapy; massage therapy
MeSH Terms: interventions — Music Therapy; Massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Music Therapy (Active Comparator): Patients randomized to the music therapy group will receive 1-3 10-40 minute music therapy sessions during each of the days of their stay on the inpatient unit. Each participant randomized to the music therapy intervention will be given a personalized CD and one portable CD player with headphones which they may keep after the study has ended.
  Interventions: Other: Music Therapy
- Massage Therapy (Active Comparator): Patients randomized to the massage therapy group will receive 1-3 10-40 minute massage treatments during each of the days of their stay on the inpatient unit.
  Interventions: Other: Massage Therapy
- Usual Care (No Intervention): The control group will continue to receive usual care while on the Family Medicine Inpatient Unit.

INTERVENTIONS:
Other: Music Therapy — Each music therapy session will begin with a brief description of the protocol, a musical introduction, a discussion of music preferences, and an informal assessment of participant needs to determine target goals, e.g., management of pain, anxiety, and other symptoms; breath control; emotional support and regulation. After the initial visit, the music therapist will create a playlist, based on participant preferences, and burn it onto a CD for the participant. The participant will be encouraged to use the book and listen to the CDs as often as he/she would like. After the initial visit, follow up visits will include techniques like music-facilitated breathing, music and imagery, music and relaxation/meditation, song writing, improvisation, singing, lyric substitution, lyric analysis, musical reminiscence, passive listening. There will be the opportunity to create music and write songs across multiple sessions, if these activities are indicated.
  Arms: Music Therapy
Other: Massage Therapy — Working with experts in hospital-based massage therapy, we have developed a semi-standardized inpatient massage protocol that utilizes Swedish techniques and acupressure. The protocol was adapted from our successful previous study of massage for perioperative care of patients undergoing implantation of permanent intravenous access devices. Massage therapists will focus on hands, feet, arms, and neck, as able, during the treatments.
  Arms: Massage Therapy

SUMMARY:
This project studies the feasibility of (1) implementing massage therapy and music therapy onto a busy medical inpatient unit at Boston Medical Center, and (2) evaluating massage therapy and music therapy's impact on patient satisfaction, patient outcomes, and cost. The investigators will conduct a randomized controlled trial comparing massage therapy, music therapy, and usual care to collect preliminary data on critical outcomes for patients (satisfaction, symptom control) and for the hospital (pain medication use and length of stay, both critical drivers of cost). The investigators anticipate using these preliminary data to apply for a future larger and longer adequately powered randomized controlled trial to definitively answer the following research questions: does implementation of an inpatient massage therapy and/or music therapy service (a) improve patient satisfaction; (b) reduce symptoms such as pain; and (c) lower health care costs through less pain medication and reduced length of stay?

DETAILED DESCRIPTION:
This randomized controlled trial compares massage therapy to usual care and music therapy to usual care for patients admitted to the Family Medicine Inpatient Unit of Boston Medical Center. Ninety family medicine inpatients will be recruited by the research assistant to participate in the study. Participants will be randomized directly following consent in a 1:1:1 ratio to massage therapy, music therapy, or usual care. Individuals assigned to the usual care group will receive the choice of a massage voucher for one massage at Boston Medical Center's Integrative Medicine program or a music therapy CD following completion of the study.

Treatment assignments will be prepared by the study biostatistician, using a permuted block method with varying block sizes of 3, 6, and 9, prior to the start of the study. These will be sealed in sequentially numbered opaque envelopes. This order will not be changed. A research assistant will take a randomization envelope, in sequential order, and read the treatment assignment to the participant following enrollment.

After enrollment and randomization is complete each day, the massage therapist and music therapist will begin to see participants for treatment. Treatments will take place in the inpatient hospital room. Curtains will be pulled closed to maintain privacy in rooms that have two beds. Both music and massage therapists will be present Monday-Sunday to provide treatment to participants.

Treatments will be attempted 1-3 times per day for the duration of the participant's stay on the unit, based on the participant's availability (they may be scheduled for diagnostic tests, imaging, consults, etc). The music and massage therapists will work down the list of participants, visiting each one by one and administering treatment (details below for each therapy). If a participant is not available at the time the therapist comes by, he/she will revisit the participant after they have gone through their list and administered treatments. Once the therapist has provided the therapy once to every patient on his/her list, he/she will begin at the top of the list and provide a second round of treatments, and repeat again for a third round as time permits.

The music therapist and massage therapist will create a note sheet each day for each participant. This will allow them to track number of treatments as well as any comments relevant to treatment (patient preferences, etc). A research assistant will collect these at the end of each day, enter them into the secure online database, and store them in a locked file cabinet.

The music therapist and massage therapist will each be given an updated list of patients to treat (first name, last initial, room number) each morning. These lists (separated by treatment group) will include the newly enrolled and randomized participants as well as those who have not yet been discharged. At the end of each day, the therapists will report to the research assistant on how many sessions were provided to each participant.

When the research assistant notes that a participant has been discharged, he/she has approximately 7 days to contact the patient (by phone or email) to administer the endline survey. Then, thirty days after discharge, the research assistant will check the participant's electronic medical record to see if he/she has been admitted again since discharge. Participants in the control group, following discharge and completion of the endline survey, will be mailed either a music/meditation CD or a voucher for massage at BMC, according to their preference.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Inpatient on the Boston Medical C enter Family Medicine inpatient service

Exclusion Criteria:

* Inability to provide informed consent
* Contagious skin disease or infection
* Hemophilia
* Thrombocytopenia
* Encephalopathy
* Dementia
* Altered mental status
* 1:1 status (requiring constant supervision)
* Any condition, as determined by the attending physician, which would prevent participation in the study.
* Observation status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-07; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction | within 7 days after discharge
  Hospital Consumer Assessment of Healthcare Providers and Systems (HCAHPS) Survey questions

SECONDARY OUTCOMES:
Pain medication use | duration of hospital stay, an expected average of 4 days
  Administration of pain medication is documented in the electronic medical record each time a dose is given. We will use the EMR to document number of doses and amount (mg) of each dose during the participant's stay.
Sedative use | duration of hospital stay, an expected average of 4 days
  Administration of sedatives is documented in the electronic medical record each time a dose is given. We will use the EMR to document number of doses and amount (mg) of each dose during the participant's stay.
Length of stay | duration of hospital stay, an expected average of 4 days
Number of re-admissions 30 days after initial discharge | 30 days post-discharge
Pain level | duration of hospital stay, an expected average of 4 days
  Pain levels are documented for every patient by nurses on a daily basis. We will utilize the electronic medical record (EMR) and document every pain evaluation (0-10 point scale of current pain intensity) performed by nurses on inpatient unit during participant's stay.

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Saper, MD, MPH, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States